CLINICAL TRIAL: NCT03617536
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of Oral CR845 in Chronic Kidney Disease Patients With Moderate-to-Severe Pruritus
Brief Title: A Study to Evaluate the Safety and Efficacy of CR845 in Chronic Kidney Disease Patients With Moderate-to-Severe Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845 210301
Record Dates: First submitted 2018-07-11; First posted 2018-08-06 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Diseases; Pruritus
Keywords: difelikefalin; CR845; Pruritus; Chronic Itch; Itch; Itching; uremic pruritus; CKD; CKD-aP; CKD-associated pruritus; Chronic Kidney Disease; Kidney dysfunction; Generalized pruritus; Hemodialysis; Dialysis; ESRD (end stage renal disease); Kidney failure, chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pruritus; Kidney Failure, Chronic | interventions — Tablets; difelikefalin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled study
Who Masked: Participant, Investigator
Masking Description: CR845 will be provided as enteric-coated tablets. All tablets are white in color with no markings and are identical in appearance, regardless of dose.
  CR845 tablets will be provided at doses of 0.25, 0.5, and 1 mg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- CR845 0.25 mg Oral Tablet (Experimental): Oral CR845 0.25 mg to be taken orally once daily for 12 weeks
  Interventions: Drug: CR845 0.25 mg Oral Tablet
- CR845 0.5 mg Oral Tablet (Experimental): Oral CR845 0.5 mg to be taken orally once daily for 12 weeks
  Interventions: Drug: CR845 0.5 mg Oral Tablet
- CR845 1 mg Oral Tablet (Experimental): Oral CR845 1 mg to be taken orally once daily for 12 weeks
  Interventions: Drug: CR845 1 mg Oral Tablet
- Placebo Oral Tablet (Placebo Comparator): Oral Placebo to be taken orally once daily
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: CR845 0.25 mg Oral Tablet — CR845 0.25 mg medication taken orally 1 time/day
  Other Names: Difelikefalin
  Arms: CR845 0.25 mg Oral Tablet
Drug: CR845 0.5 mg Oral Tablet — CR845 0.5 mg medication taken orally 1 time/day
  Other Names: Difelikefalin
  Arms: CR845 0.5 mg Oral Tablet
Drug: CR845 1 mg Oral Tablet — CR845 1 mg medication taken orally 1 time/day
  Other Names: Difelikefalin
  Arms: CR845 1 mg Oral Tablet
Drug: Placebo Oral Tablet — Placebo tablet taken orally 1 time/day
  Arms: Placebo Oral Tablet

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of 3 dose levels of oral CR845 compared to placebo in reducing the intensity of itch in chronic kidney disease (CKD) patients with moderate-to-severe pruritus. This study will consist of a Screening Period, a 7-day Run-in Period, a 12 week Treatment Period, and a Follow-up Visit (approximately 7 days after the last dose of study drug).

DETAILED DESCRIPTION:
This study will consist of a Screening Period, a 7-day Run-in Period, a 12 week Treatment Period, and a Follow-up Visit (approximately 7 to 10 days after the last dose of study drug). Informed consent will be obtained prior to performing any study-specific procedures. Screening will occur within 7 to 28 days prior to randomization to assess eligibility.

If patients continue to meet all inclusion and no exclusion criteria at the end of the 7-day Run-in Period, they will be randomized in a 1:1:1:1 ratio to receive orally once daily either placebo or CR845 tablets at doses of 0.25, 0.5 or 1 mg. Randomization will be stratified according to the patient's renal disease status: moderate CKD; severe CKD non-dialysis; severe CKD on dialysis (ie, 3 categories). A final safety Follow-up Visit will be conducted 7 to 10 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into the study, a patient must meet the following criteria:

* CKD patients with stage III, IV, or V (ie, moderate renal impairment with estimated glomerular filtration rate (GFR) ≥30 and <60 mL/min/1.73 m2 or severe renal impairment with estimated GFR <30 mL/min/1.73 m2).
* For severe CKD patients on hemodialysis, they must be receiving hemodialysis 3 times per week for at least 3 months prior to the start of screening;
* Prior to randomization:

  1. Has completed at least 4 Worst Itching Intensity NRS worksheets from the start of the 7-day Run-in Period;
  2. Has a mean baseline Worst Itching Intensity NRS score ≥5, defined as the average of all non-missing scores reported from the start of the 7-day Run-in Period.

Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

* Patients not currently on dialysis who are likely to initiate routine dialysis during study participation;
* Scheduled to receive a kidney transplant during the study;
* New or change of treatment received for itch including antihistamines and corticosteroids (oral, intravenous [IV], or topical) within 14 days prior to screening;
* Received another investigational drug within 30 days prior to the start of screening or is planning to participate in another clinical study while enrolled in this study;
* Received ultraviolet B treatment within 30 days prior to the start of screening or anticipates receiving such treatment during the study;
* Participated in a previous clinical study with CR845.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Menzaghi, PhD, Study Director — Cara Therapeutics
Locations (58):
- United States (58):
  - Cara Therapeutics Study Site, Birmingham, Alabama
  - Cara Therapeutics Study Site, Florence, Alabama
  - Cara Therapeutics Study Site, Phoenix, Arizona
  - Cara Therapeutics Study Site, Prescott, Arizona
  - Cara Therapeutics Study Site, Sun City, Arizona
  - Cara Therapeutics Study Site, Harrisburg, Arkansas
  - Cara Therapeutics Study Site, Bakersfield, California
  - Cara Therapeutics Study Site 2, Bakersfield, California
  - Cara Therapeutics Study Site, Canyon Country, California
  - Cara Therapeutics Study Site, Escondido, California
  - Cara Therapeutics Study Site, Lomita, California
  - Cara Therapeutics Study Site, Northridge, California
  - Cara Therapeutics Study Site, Riverside, California
  - Cara Therapeutics Study Site, Sacramento, California
  - Cara Therapeutics Study Site, Whittier, California
  - Cara Therapeutics Study Site, Denver, Colorado
  - Cara Therapeutics Study Site, Washington D.C., District of Columbia
  - Cara Therapeutics Study Site, Edgewater, Florida
  - Cara Therapeutics Study Site, Hialeah, Florida
  - Cara Therapeutics Study Site, Hollywood, Florida
  - Cara Therapeutics Study Site, Lake Worth, Florida
  - Cara Therapeutics Study Site 1, Miami, Florida
  - Cara Therapeutics Study Site 2, Miami, Florida
  - Cara Therapeutics Study Site, Ocala, Florida
  - Cara Therapeutics Study Site, Orlando, Florida
  - Cara Therapeutics Study Site, Tampa, Florida
  - Cara Therapeutics Study Site, Temple Terrace, Florida
  - Cara Therapeutics Study Site, Augusta, Georgia
  - Cara Therapeutics Study Site, Sandy Springs, Georgia
  - Cara Therapeutics Study Site, Crystal Lake, Illinois
  - Cara Therapeutics Study Site, Evanston, Illinois
  - Cara Therapeutics Study Site, Iowa City, Iowa
  - Cara Therapeutics Study Site, Metairie, Louisiana
  - Cara Therapeutics Study Site, New Orleans, Louisiana
  - Cara Therapeutics Study Site, Zachary, Louisiana
  - Cara Therapeutics Study Site, Baltimore, Maryland
  - Cara Therapeutics Study Site, Takoma Park, Maryland
  - Cara Therapeutics Study Site, Flint, Michigan
  - Cara Therapeutics Study Site 2, Flint, Michigan
  - Cara Therapeutics Study Site, Roseville, Michigan
  - Cara Therapeutics Study Site, Saint Clair, Michigan
  - Cara Therapeutics Study Site, Kansas City, Missouri
  - Cara Therapeutics Study Site, Brooklyn, New York
  - Cara Therapeutics Study Site, Mineola, New York
  - Cara Therapeutics Study Site, Rocky Mount, North Carolina
  - Cara Therapeutics Study Site, Columbus, Ohio
  - Cara Therapeutics Study Site, Norman, Oklahoma
  - Cara Therapeutics Study Site, Camp Hill, Pennsylvania
  - Cara Therapeutics Study Site, Providence, Rhode Island
  - Cara Therapeutics Study Site, Warwick, Rhode Island
  - Cara Therapeutics Study Site, Greenville, South Carolina
  - Cara Therapeutics Study Site, Rapid City, South Dakota
  - Cara Therapeutics Study Site, Corsicana, Texas
  - Cara Therapeutics Study Site, Gonzales, Texas
  - Cara Therapeutics Study Site, Houston, Texas
  - Cara Therapeutics Study Site, Plano, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CR845 0.25 mg Oral Tablet | CR845 0.5 mg Oral Tablet | CR845 1 mg Oral Tablet | Placebo Oral Tablet
Started | 69 | 66 | 67 | 67
Completed | 60 | 57 | 54 | 57
Not Completed | 9 | 9 | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CR845 0.25 mg Oral Tablet | CR845 0.5 mg Oral Tablet | CR845 1 mg Oral Tablet | Placebo Oral Tablet | Total
Number analyzed (Participants) | 69 | 66 | 67 | 67 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (11.0) | 69.0 (12.0) | 67.5 (10.7) | 65.6 (12.1) | 66.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 32 | 30 | 130
  Male | 34 | 33 | 35 | 37 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 5 | 4 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 2
  Black or African American | 17 | 12 | 15 | 17 | 61
  White | 49 | 49 | 48 | 47 | 193
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Mean of the Daily 24-hour Worst Itching Intensity Numerical Rating Scale (NRS) Score During Week 12
Description: Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable". Higher scores meant worse itch intensity.
Time Frame: Baseline, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CR845 0.25 mg Oral Tablet | CR845 0.5 mg Oral Tablet | CR845 1 mg Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 69 | 66 | 67 | 67
score on a scale | -3.99 [-4.62 to -3.36] | -3.84 [-4.50 to -3.18] | -4.42 [-5.08 to -3.76] | -3.32 [-3.97 to -2.68]

2. Secondary Outcome: Change From Baseline in Total Skindex-10 Scale Score at the End of Week 12
Description: The Skindex-10 Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past week. The questions cover 3 domains: disease, mood/emotional distress, and social functioning domain. The Skindex-10 has 10 questions; the total Skindex-10 score ranges from 0 to 60. A lower total score represents better quality of life.
Time Frame: Baseline, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CR845 0.25 mg Oral Tablet | CR845 0.5 mg Oral Tablet | CR845 1 mg Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 69 | 66 | 67 | 67
score on a scale | -21.19 [-24.34 to -18.04] | -22.13 [-25.37 to -18.89] | -23.57 [-27.00 to -20.14] | -19.95 [-23.17 to -16.73]

3. Secondary Outcome: Change From Baseline in 5-D Itch Scale Score at the End of Week 12
Description: The 5-D Itch Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past 2 weeks. The questions cover five dimensions of itch including the degree, duration of itch/day, direction (improvement/worsening), disability (impact on activities such as work), and body distribution of itch. The 5-D Itch Scale has 5 questions; the total 5-D Itch Scale score ranges from 5 to 25, with higher scores indicating worse responses.
Time Frame: Baseline, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CR845 0.25 mg Oral Tablet | CR845 0.5 mg Oral Tablet | CR845 1 mg Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 69 | 66 | 67 | 67
score on a scale | -6.17 [-7.10 to -5.25] | -6.84 [-7.78 to -5.90] | -6.97 [-7.97 to -5.97] | -5.74 [-6.69 to -4.80]

4. Secondary Outcome: Reduction of Itch Intensity as Assessed by the Proportion of Patients Achieving an Improvement From Baseline ≥3 Points With Respect to the Weekly Mean of the Daily 24-hour Worst Itching Intensity NRS Score at Week 12
Time Frame: Week 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | CR845 0.25 mg Oral Tablet | CR845 0.5 mg Oral Tablet | CR845 1 mg Oral Tablet | Placebo Oral Tablet
Number analyzed (Participants) | 69 | 66 | 67 | 67
percentage of subjects | 66.2 [53.00 to 77.32] | 64.8 [51.18 to 76.30] | 72.1 [58.62 to 82.45] | 57.9 [44.15 to 70.49]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded starting at the Screening Visit and continuing through the Follow-up Visit (7 to 10 days after the last dose of study drug).
Arm/Group | CR845 0.25 mg Oral Tablet | CR845 0.5 mg Oral Tablet | CR845 1 mg Oral Tablet | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/66 | 1/67 | 3/67
Serious Adverse Events (participants affected / at risk) | 9/69 | 9/66 | 9/67 | 5/67
Other Adverse Events (participants affected / at risk) | 12/69 | 10/66 | 15/67 | 8/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 0.25 mg Oral Tablet (N=69) | CR845 0.5 mg Oral Tablet (N=66) | CR845 1 mg Oral Tablet (N=67) | Placebo Oral Tablet (N=67)
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Athenia (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 0.25 mg Oral Tablet (N=69) | CR845 0.5 mg Oral Tablet (N=66) | CR845 1 mg Oral Tablet (N=67) | Placebo Oral Tablet (N=67)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 4
Fatigue (General disorders) | 4 | 1 | 3 | 1
Hypertension (Vascular disorders) | 4 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 4 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT03617536/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT03617536/SAP_001.pdf